CLINICAL TRIAL: NCT06563934
Title: A Randomized Controlled Trial Evaluating the Effects of Oral Enterobacterial Capsules in Liver Cancer Patients Treated With Tyrosine Kinase Inhibitors (TKIs) in Combination With Immune Checkpoint Inhibitors (ICIs)
Brief Title: Gut Microbiota in Liver Cancer (Treated With TKIs In Combination With ICIs)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xu Yong, MD (Other)
Collaborators: Nanjing Xiershou Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Xu Yong, MD, Secretary of the Party Committee, Shenzhen Third People's Hospital
Organization: Shenzhen Third People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY2024-177
Record Dates: First submitted 2024-08-13; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, randomized, double-blind controlled trial. The clinical study is divided into 2 groups: Group 1) Patients in the control group were given lenvatinib 8mg (≤ 60 kg body weight) or 12 mg (> 60 kg body weight) orally once a day, combined with PD-1 monoclonal antibody 200mg intravenously once every 3 weeks until disease progression, intolerable toxicity or death, and patients in the control group were given intestinal bacteria capsules placebo. Group 2) Patients in the study group were given lenvatinib 8 mg (≤ 60 kg body weight) or 12 mg (> 60 kg body weight) orally once a day in combination with PD-1 monoclonal antibody 200 mg intravenously every 3 weeks until disease progression, intolerable toxicity, or death, and patients in this study group were given intestinal bacteria capsules.
Who Masked: Participant, Investigator
Masking Description: This is a prospective, single-center, randomized, double-blind controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Lenvatinib + PD-1 monoclonal antibody + Enterobacterium capsules (Experimental): 1. Lenvatinib 8mg (≤60 kg body weight) or 12 mg (> 60 kg body weight) orally once a day. PD-1 monoclonal antibody 200mg i.v. once every 3 weeks.
  2. Enterobacterium capsules (300 mg/per capsule) orally 6 capsules/day for 10 consecutive days, and then discontinued to the next course of treatment.
  Interventions: Biological: Oral enterobacterium capsules; Drug: Lenvatinib + PD-1 monoclonal antibody
- Lenvatinib + PD-1 monoclonal antibody + Enterobacterium capsules placebo (Placebo Comparator): 1. Lenvatinib 8mg (≤60 kg body weight) or 12 mg (> 60 kg body weight) orally once a day. PD-1 monoclonal antibody 200mg i.v. once every 3 weeks.
  2. Enterobacterium capsules placebo (300 mg/per capsule) orally 6 capsules/day for 10 consecutive days, and then discontinued to the next course of treatment.
  Interventions: Drug: Lenvatinib + PD-1 monoclonal antibody; Biological: Oral enterobacterium capsules placebo

INTERVENTIONS:
Biological: Oral enterobacterium capsules — Enterobacterium capsules (300 mg/per capsule) orally 6 capsules/day for 10 consecutive days.
  Arms: Experimental: Lenvatinib + PD-1 monoclonal antibody + Enterobacterium capsules
Drug: Lenvatinib + PD-1 monoclonal antibody — Lenvatinib 8mg (≤60 kg body weight) or 12 mg (> 60 kg body weight) orally once a day.
  PD-1 monoclonal antibody 200mg i.v. once every 3 weeks.
Biological: Oral enterobacterium capsules placebo — Enterobacterium capsules placebo (300 mg/per capsule) orally 6 capsules/day for 10 consecutive days.
  Arms: Lenvatinib + PD-1 monoclonal antibody + Enterobacterium capsules placebo

SUMMARY:
To evaluate the additional efficacy and safety of oral enterobacterial capsules in patients with intermediate and advanced liver cancer and treated with tyrosine kinase inhibitors (TKIs) combined with immunotherapy.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, double-blind controlled trial. The clinical study is divided into 2 groups:

Group 1) Patients in the control group were given lenvatinib 8mg (≤ 60 kg body weight) or 12 mg (> 60 kg body weight) orally once a day, combined with PD-1 monoclonal antibody 200mg intravenously once every 3 weeks until disease progression, intolerable toxicity or death, and patients in the control group were given intestinal bacteria capsules placebo.

Group 2) Patients in the study group were given lenvatinib 8 mg (≤ 60 kg body weight) or 12 mg (> 60 kg body weight) orally once a day in combination with PD-1 monoclonal antibody 200 mg intravenously every 3 weeks until disease progression, intolerable toxicity, or death, and patients in this study group were given intestinal bacteria capsules.

Oral administration of intestinal bacteria capsules 6 capsules/day, after observing no adverse reactions, oral administration for 10 consecutive days, 6 capsules/day from the second day to the tenth day, and then discontinued to the next course of treatment.

Total course of treatment: a total of 4 courses of oral intestinal bacteria capsules, each course of oral administration for 10 days, and a course of 21 days; A course of TKI combined with immune checkpoint inhibitors treatment is 21 days until the disease progresses or intolerable toxicity and side effects appear.

Observe the metrics: Primary Clinical Endpoint - Progression-Free Survival (PFS); Secondary Clinical Endpoints - Overall Growth Phase (OS), Objective Response Rate (ORR), Duration of Response (DOR), and Disease Control Rate (DCR). The new RECIST1.1 criteria were used for the efficacy evaluation system, the CTCAE5.0 grading system was used for the evaluation of common adverse reactions during treatment, and other indicators included imaging including conventional biochemical indexes such as CT and ultrasound, as well as quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. Confirmed imaging or histological diagnosis of unresectable HCC, BCLC stadium B or C;
3. Previous treatment without systemic therapy;
4. Intended to be treated with anti-angiogenic targeted drugs combined with immune checkpoint inhibitors;
5. Child-Pugh Grade A;
6. ≥ 1 measurable lesion (RECIST v1.1)
7. ECOG PS 0-1

Exclusion Criteria:

1. Usage of antibiotics within 2 weeks prior enrollment;
2. Diagnosis of immunodeficiency (e.g. HIV, immunosuppressants)
3. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
4. Female patients who are pregnant or breastfeeding;
5. Patients with untreated acute or chronic active hepatitis B or hepatitis C infection.
6. Those who are currently undergoing clinical trials of other drugs;
7. Other patients who are considered by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Objective Progression-Free Survival (PFS) | Up to approximately 1 years
  To analyse the Progression-Free Survival (PFS) of patients
Objective Secondary Clinical Endpoints - Overall Growth Phase (OS) | Up to approximately 1 years
  To analyse the Secondary Clinical Endpoints - Overall Growth Phase (OS) of patients
Objective Objective Response Rate (ORR) | Up to approximately 1 years
  To exprole the Objective Response Rate (ORR) of patients
ObjectiveDuration of Response (DOR) | Up to approximately 1 years
  To analyse the Duration of Response (DOR) of patients
Diversity analysis | Up to approximately 1 years
  We will use 16S rRNA sequencing to measure fecal sample. The alpha and beta diversity of gut microbiota will be analyzed, including a series of statistical analysis indexes such as Chao, Shannon, Simpsonace, Simpson and Coverage, in order to reflect the microbial community diversity.
Species differential analysis | Up to approximately 1 years
  We will use 16S rRNA sequencing to measure fecal sample. Based on the results of species annotation, the PCA、PCoA and NMDS analysis will be used to assess the similarities and differences in species composition.
Feces Metabolomics | Up to approximately 1 years
  Changes of metabolites in feces measured by metabolomic mass spectrometry, unsupervised PCA (principal component analysis) was performed by statistics function prcomp, identified metabolites were annotated using KEGG Compound database.
Serum Metabolomics | Up to approximately 1 years
  Changes of metabolites in serum measured by metabolomic mass spectrometry, unsupervised PCA (principal component analysis) was performed by statistics function prcomp, identified metabolites were annotated using KEGG Compound database.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Xu, Dr, Principal Investigator — Secretary of the Party Committee of the Shenzhen Third People's Hospital

IPD SHARING:
Plan to Share IPD: No